CLINICAL TRIAL: NCT04482374
Title: Effects of Puberty and Pubertal Suppression on Insulin Sensitivity, Metabolic Rate and Vascular Health
Brief Title: Puberty Suppression and Cardiometabolic Health
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-2109
Record Dates: First submitted 2020-06-30; First posted 2020-07-22 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Transgenderism; Insulin Sensitivity/Resistance; Endothelial Dysfunction; Vascular Stiffness
MeSH Terms: conditions — Transsexualism; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender females: Transgender females who plan to start a gonadotropin releasing hormone agonist clinically in the next 2 months
- Cisgender males: Cisgender male controls

SUMMARY:
This observational study will evaluate the effect of puberty suppression on insulin sensitivity, metabolic rate and vascular health among transgender female youth at baseline and 6 months after initiation of a gondoatropin releasing hormone agonist compared to matched cisgender male controls.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a transgender female or cisgender male
* Age 9-14 years at the time of enrollment
* Tanner Stage 2-3 baseline pubertal development
* Plan to start gonadotropin releasing hormone analogue clinically in < 2 months (for transgender females only)

Exclusion Criteria:

* Cognitive, psychiatric, or physical impairment resulting in inability to tolerate the study procedures
* Type 1 or 2 diabetes (by medical history)
* On any medications that affect insulin sensitivity (e.g. metformin, antipsychotics)
* Hypertension (resting BP ≥ 140/90 mm/Hg)
* Weight > 400 lbs
* On estrogen- or progesterone-containing medications at baseline
* >3 hours of moderate-to-vigorous physical activity on the 3DPAR at the screening visit

Ages: 9 Years to 14 Years | Sex: Male
Age Groups: Child
Gender Based: Yes — Transgender females, cisgender males
Study Population: 15 transgender females (male sex assigned at birth, female gender identity) and 15 cisgender males
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Baseline, 6 months
  Insulin sensitivity assessed by the oral minimal model

SECONDARY OUTCOMES:
Change in body composition (fat mass, fat-free mass) | Baseline, 6 months
  Body composition measured by DXA
Change in resting metabolic rate | Baseline, 6 months
  Resting metabolic rate assessed by indirect calorimetry
Change in endothelial function | Baseline, 6 months
  Endothelial function assessed by brachial artery flow mediated dilation
Change in large elastic artery stiffness | Baseline, 6 months
  Large elastic assessed by carotid ultrasound
Change in cerebrovascular function | Baseline, 6 months
  Middle cerebral artery blood flow assessed using bilateral transcranial Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Natalie J Nokoff, MD, MSCS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided